CLINICAL TRIAL: NCT06254443
Title: Comparison of Oral Polyethylene Glycol and Enema for Diagnostic Efficacy in Urgent Colonoscopy for Acute Lower Gastrointestinal Bleeding: a Multicenter, Randomized, Non-inferiority Trial
Brief Title: Oral PEG vs. Enema in Urgent Colonoscopy for ALGIB
Acronym: CANDLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Min Li, Deputy Director of Science and Technology Department, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BFHHZML20240002
Record Dates: First submitted 2024-01-07; First posted 2024-02-12 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Acute Lower Gastrointestinal Bleeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral PEG group (Other): Following the administration protocol recommended by the Chinese expert consensus for PEG, a 3 L PEG regimen is employed. The regimen involves segmented intake, with 1 L taken 10-12 hours before the intestinal examination and an additional 2 L taken 4-6 hours before the examination on the day of the procedure.
  Interventions: Other: PEG Bowel preparation
- Enema group (Other): Enema is administered using either normal saline or 1% soapy water for cleansing until the effluent is clear of fecal debris, or until a total volume of 3000 ml of enema solution has been administered. The enema should be initiated 4-6 hours before colonoscopy, with the dosage and frequency of incremental enemas determined based on the patient's tolerance. The final enema administration should be completed no later than 10 minutes before the scheduled colonoscopy.
  Interventions: Other: Enema Bowel preparation

INTERVENTIONS:
Other: Enema Bowel preparation — Enema Group (Experimental Group): Enema is administered using either normal saline or 1% soapy water for cleansing until the effluent is clear of fecal debris, or until a total volume of 3000 ml of enema solution has been administered. The enema should be initiated 4-6 hours before colonoscopy, with the dosage and frequency of incremental enemas determined based on the patient's tolerance. The final enema administration should be completed no later than 10 minutes before the scheduled colonoscopy.
  Arms: Enema group
Other: PEG Bowel preparation — Oral PEG Group (Control Group): Following the administration protocol recommended by the Chinese expert consensus for PEG, a 3 L PEG regimen is employed. The regimen involves segmented intake, with 1 L taken 10-12 hours before the intestinal examination and an additional 2 L taken 4-6 hours before the examination on the day of the procedure.
  Arms: Oral PEG group

SUMMARY:
The main goal of this study is to assess whether the diagnostic efficacy of enema is non-inferior to that of oral polyethylene glycol (PEG) in acute lower gastrointestinal bleeding (ALGIB) patients requiring urgent colonoscopy. The secondary objectives include: 1) evaluating potential differences between the enema and oral PEG groups in terms of the difficulty and safety of colonoscopy, as well as exacerbation of bleeding; 2) conducting subgroup analyses to compare the effectiveness of the two bowel preparation methods in specific populations, exploring potential candidate groups for different bowel preparation strategies, and promoting individualized diagnosis and treatment for ALGIB.

DETAILED DESCRIPTION:
This is a multicenter, prospective, single-blind, randomized controlled, non-inferiority study. The study includes the following steps:

Step 1: Participants will be enrolled based on predefined criteria, and demographic data, fasting water duration, accompanying symptoms, smoking history, alcohol consumption history, antithrombotic drug usage, previous history of lower gastrointestinal bleeding, Charlson comorbidity index, vital signs at admission, and laboratory results at admission will be collected.

Step 2: All participants will undergo stratified block randomization, and based on the randomization results, participants will receive bowel preparation using either PEG or enema. Subsequently, all participants will undergo urgent colonoscopy within 48 hours from admission.

Step 3: Follow-up records will be conducted at the following time points:

1. Before colonoscopy:

   * Record the specific method and dosage of actual bowel preparation.
   * Record changes in vital signs, symptoms, and signs before and after bowel preparation, as well as occurrences of adverse events.
   * Conduct a satisfaction survey of bowel preparation.
2. During colonoscopy:

   - Record patient pain scores, Boston bowel preparation scores, cecal intubation time, lesion detection time, total procedure time, maximum insertion depth, observation of active bleeding, endoscopic diagnosis, endoscopic hemostasis, and perforation.
3. After colonoscopy:

   * Record postoperative adverse events, need for repeat endoscopy, transfusion, intervention or surgery, and final discharge diagnosis.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting with hematochezia who were admitted to our hospitals were eligible for the study. Patients were included if they met the following criteria:

1. Had the last bloody bowel movement within 24 hours of presentation;
2. Aged 18 years or over
3. Had indications for clinical colonoscopy

Exclusion Criteria:

1. Known or suspected upper gastrointestinal bleeding meeting any of the following criteria:

   A. Presence of hematemesis or black vomiting. B. Bloody or coffee nasogastric aspirate. C. Endoscopic evidence of acute upper gastrointestinal bleeding, such as gastric or duodenal ulcer bleeding, esophagogastric variceal bleeding, etc.
2. Previous colonoscopy has been performed at an external institution with a confirmed diagnosis.
3. Presence of primary or secondary coagulation disorders.
4. History of bowel diversion surgery (including partial colon resection).
5. Hemodynamic instability persists after fluid resuscitation (shock index greater than 1).
6. Interventional treatment has been performed and hemostasis has been successfully achieved.
7. Requires transfer to an intensive care unit due to the severity of the condition.
8. Unable to comply with oral polyethylene glycol administration or enema procedures.
9. Known or suspected relative contraindications to colonoscopy, such as toxic megacolon, acute intestinal obstruction, acute myocardial infarction, heart failure, severe liver failure, and end-stage renal disease.
10. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Endoscopic diagnosis rate | During the colonoscopy (up to 48 hours from admission)
  Including the definite diagnosis and presumptive diagnosis

SECONDARY OUTCOMES:
Cecal intubation time | During the colonoscopy (up to 48 hours from admission)
  The duration from the insertion of the colonoscope through the anus to reaching the cecum.
Lesion detection time | During the colonoscopy (up to 48 hours from admission)
  The duration from the insertion of the colonoscope through the anus to the initial identification of lesions.
Total procedure time | During the colonoscopy (up to 48 hours from admission)
  The duration from the insertion of the colonoscope through the anus to the withdrawal from the anus.
Cecal intubation rate | During the colonoscopy (up to 48 hours from admission)
  The proportion of patients in the study group in whom successful cecal intubation was achieved, relative to the total number of patients in the group.
Rate of bowel preparation related adverse events | From the start of bowel preparation to the end of bowel preparation (assessed up to 44 hours from admission)
  Bowel preparation related adverse events included nausea, vomiting, bloating, hypotension, heart failure, electrolyte imbalance, aspiration pneumonia, etc.
Rate of colonoscopy related adverse events | From the start of colonoscopy to the time of discharge (assessed up to 72 hours from admission)
  Colonoscopy related adverse events included perforation, recurrent bleeding, post-operational infection and death.
Rate of patients who sufferred from exacerbation of ALGIB | From the start of bowel preparation to the end of bowel preparation (assessed up to 44 hours from admission)
  Exacerbation of ALGIB was defined as patients' subjective bleeding symptoms were worse than before the start of bowel preparation, or patients had a decrease in hemoglobin of more than 2g/L before and after bowel preparation.
Bowel preparation satisfaction score | At the end of bowel preparation (assessed up to 48 hours from admission)
  The satisfaction score of bowel preparation was evaluated from three dimensions: mood, discomfort symptoms, and general feeling, with each dimension ranging from 0 to 5 indicating from the worst to the best.
Boston bowel preparation score | During the colonoscopy (up to 48 hours from admission)
  A score of 0 to 9 on the Boston Bowel Preparation scale indicates worst to best.
Endoscopic hemostasis rate | During the colonoscopy (up to 48 hours from admission)
  The rate of performance of endoscopic hemostasis.
Intervention or surgery rate | From the end of colonoscopy to the time of discharge (assessed up to 72 hours from admission)
  The rate of patients who underwent angiographic therapy or surgery after the primary colonoscopy.
Repeated endoscopy rate | From the end of colonoscopy to the time of discharge (assessed up to 72 hours from admission)
  The rate of patients who received a second-look of colonoscopy after the primary colonoscopy.
Transfusion rate | From the end of colonoscopy to the time of discharge (assessed up to 72 hours from admission)
  The rate of patients who need red blood cell transfusion after the primary colonoscopy.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Tongliao City Hospital, Tongliao, Neimenggu
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Beijing Friendship Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No